CLINICAL TRIAL: NCT04512898
Title: Effect of Helicobacter Pylori Eradication on Symptoms and Quality of Life of Irritable Bowel Syndrome: A Prospective Study
Brief Title: Helicobacter Pylori Eradication and Irritable Bowel Syndrome: A Prospective Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidi Karam, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H. Pylori
Record Dates: First submitted 2020-08-03; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Patients with IBS and have H. pylori
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with IBS (Experimental): Patients with IBS and positive H. pylori.
  Interventions: Drug: Triple therapy for H.pylori

INTERVENTIONS:
Drug: Triple therapy for H.pylori — Triple therapy of proton pump inhibitors, clarithromycin and metronidazole.

SUMMARY:
H. Pylori is frequently observed in patients with irritable bowel syndrome(IBS). However, the effect of H. pylori eradication on IBS is not clear.

DETAILED DESCRIPTION:
Patients with IBS symptoms using Rome IV criteria will be included. Testing for H. pylori will be done. Patients with H. pylori will receive triple therapy and followed after two weeks for eradication and assessment of IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with IBS and H.pylori

Exclusion Criteria:

* Patients received previous treatment of H.pylori
* Patients receiving treatment for IBS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-10 (Estimated); Primary Completion 2020-11-10 (Estimated); Study Completion 2020-11-10 (Estimated)

PRIMARY OUTCOMES:
Questionnaire for Rome IV criteria | 2 weeks
  Symptoms of IBS

SECONDARY OUTCOMES:
Quality of life questionnaire | 2 weeks
  Quality of life.

IPD SHARING:
Plan to Share IPD: No